CLINICAL TRIAL: NCT01344018
Title: A Phase III Randomized Study of Preoperative Radiotherapy Plus Surgery Versus Surgery Alone for Patients With Retroperitoneal Sarcoma (RPS)
Brief Title: Surgery With or Without Radiation Therapy in Untreated Nonmetastatic Retroperitoneal Sarcoma
Acronym: STRASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62092-22092; EORTC-62092 (Other: EORTC); EORTC-22092 (Other: EORTC); EU-21113 (Other: EU)
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult malignant fibrous histiocytoma; adult malignant mesenchymoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Malignant mesenchymal tumor | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery alone (Active Comparator): En-bloc resection of surrounding tissues and organs when located within 1 to 2 cm from the surface tumor, even when not infiltrated.
  Interventions: Procedure: therapeutic conventional surgery
- Preoperative radiotherapy followed by en-bloc surgery (Experimental): 3D-CRT or IMRT to a dose of 50.4 Gy/28 daily fractions
  Interventions: Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Procedure: therapeutic conventional surgery
Radiation: 3-dimensional conformal radiation therapy
  Arms: Preoperative radiotherapy followed by en-bloc surgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether surgery is more effective with or without radiation therapy in treating nonmetastatic retroperitoneal soft tissue sarcoma.

PURPOSE: This randomized phase III trial is studying radiation therapy followed by surgery to see how well it works compared with surgery alone in treating patients with previously untreated nonmetastatic retroperitoneal soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether there is a difference in abdominal recurrence-free survival between retroperitoneal soft tissue sarcoma patients undergoing curative intent surgery alone and those undergoing preoperative radiotherapy followed by curative-intent surgery.

Secondary

* To assess whether there is a difference in metastasis-free survival, abdominal recurrence-free interval, and overall survival between these patients.
* To assess tumor response in patients undergoing preoperative radiotherapy.
* To assess toxicity of preoperative radiotherapy given prior to curative-intent surgery in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to institution and WHO performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo surgical resection of the tumor mass within 4 weeks following randomization.
* Arm II: Patients undergo 3-dimensional conformal radiation therapy (RT) or intensity-modulated RT within 8 weeks after randomization. RT continues 5 days a week for approximately 5.5 weeks. Patients undergo surgical resection of the tumor mass within 4-8 weeks after the completion of RT.

Tumor tissue, normal abdominal wall fat, and peripheral blood may be collected during surgery to identify new prognostic factors for translational research.

After completion of study therapy, patients are followed at day 60 post-surgery and every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed retroperitoneal sarcoma (RPS) by local pathologist, imaging-guided or surgical biopsy, including the following:

  * Primary soft tissue sarcoma of retroperitoneal space or infra-peritoneal spaces of pelvis
  * Sarcoma not originated from bone structure, abdominal, or gynecological viscera
  * Unifocal tumor (not multifocal disease)
  * Absence of extension through the sciatic notch or across the diaphragm
* The following histological sub-types are not allowed:

  * Gastrointestinal stromal tumor (GIST)
  * Rhabdomyosarcomas
  * Primitive neuroectodermal tumor (PNET) or other small round blue cells sarcoma
  * Osteosarcoma or chondrosarcoma
  * Aggressive fibromatosis
  * Sarcomatoid or metastatic carcinoma
* No metastatic disease
* Untreated disease
* Tumor must be operable and suitable for radiotherapy, based on the following criteria:

  * Pre-treatment CT scan/MRI and multidisciplinary consultation with surgeon, radiation oncologist, and radiologist (anticipated macroscopically complete resection, R0/R1 resection)

    * No surgery anticipated to be R2 on the CT scan before randomization
  * Must have American Society of Anesthesiologist (ASA) score ≤ 2
  * None of the following unresectable criteria:

    * Involvement of superior mesenteric artery
    * Involvement of aorta
    * Involvement of bone
* Must have radiologically measurable disease (RECIST 1.1), as confirmed by abdomino-pelvic CT (with IV and PO contrast) or MRI (with IV contrast)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* WBC ≥ 2,500/mm^3
* Platelet count ≥ 80,000/mm^3
* Total bilirubin < 1.5 times the upper limit normal
* Calculated creatinine clearance normal
* Functional contra-lateral kidney to the side involved by the RPS as assessed by intravenous pyelogram
* Adequate cardiac function (NYHA class I-II)
* ECG normal (without clinically significant abnormalities)
* No history of any of the following disorders:

  * Bowel obstruction
  * Mesenteric ischemia
  * Severe chronic inflammatory bowel disease
* Negative pregnancy test
* Not pregnant or nursing concurrently and for at least 1 month after the surgery
* Fertile patients must use effective contraception during the study treatment period and for at least 1 month after the surgery
* No co-existing malignancy within the past 5 years, except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior surgery (excluding diagnosis biopsy), radiotherapy, or systemic therapy
* No prior abdominal or pelvic irradiation for another prior malignancy or other disease
* No concurrent systemic anticancer treatment (chemotherapy, molecular-targeted therapy)
* No postoperative radiotherapy planned

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bonvalot, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Rick LM Haas, MD, Study Chair — The Netherlands Cancer Institute
Locations (37):
- Dana-Farber Cancer Institute & Harvard Medical School, Boston, Massachusetts, United States
- Belgium (2):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet (101), Brussels
  - U.Z. Gasthuisberg, Leuven
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Université de Montreal - Hopital Notre-Dame, Montreal Quebec, Quebec
- University Copenhagen, Herlev, Denmark
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Universitaetsklinikum, Cologne
  - UniversitaetsMedizin Mannheim, Mannheim
  - Klinikum der Universitaet, München
  - Technische Universitaet Muenchen, München
- Italy (4):
  - Centro Di Riferimento Oncologico, Aviano
  - Istituto Clinico Humanitas, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto, Padua
- Netherlands (4):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Radboud University Medical Center, Nijmegen
- Radium Hospitalet, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Center, Warsaw, Poland
- Spain (2):
  - Hospital General Vall d'Hebron, Barcelona
  - Hospital Universitario San Carlos, Madrid
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (11):
  - Queen Elizabeth Medical Center, Birmingham
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - General Western Hospital, Edinburgh
  - Beatson-Gartnavel General Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St. James'S University Hospital, Leeds
  - University College Hospital, London
  - Royal Marsden Hospital - Chelsea, London, London
  - Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle
  - Nottingham University Hospitals NHS Trust - City Hospital campus, Nottingham
  - Weston Park Hospital, Sheffield

REFERENCES:
- [Derived] Bonvalot S, Gronchi A, Le Pechoux C, Swallow CJ, Strauss D, Meeus P, van Coevorden F, Stoldt S, Stoeckle E, Rutkowski P, Rastrelli M, Raut CP, Hompes D, De Paoli A, Sangalli C, Honore C, Chung P, Miah A, Blay JY, Fiore M, Stelmes JJ, Dei Tos AP, Baldini EH, Litiere S, Marreaud S, Gelderblom H, Haas RL. Preoperative radiotherapy plus surgery versus surgery alone for patients with primary retroperitoneal sarcoma (EORTC-62092: STRASS): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2020 Oct;21(10):1366-1377. doi: 10.1016/S1470-2045(20)30446-0. Epub 2020 Sep 14. PMID 32941794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 266 (216 by EORTC members and 50 by non-EORTC members) patients were registered by 30 institutions between January 18, 2012 and April 10, 2017.
Groups:
- Surgery Alone: En-bloc resection of surrounding tissues and organs when located within 1 to 2 cm from the surface tumor, even when not infiltrated.
  therapeutic conventional surgery
- Preoperative Radiotherapy Followed by En-bloc Surgery: 3D-CRT or IMRT to a dose of 50.4 Gy/28 daily fractions
  therapeutic conventional surgery
  3-dimensional conformal radiation therapy
Period: Overall Study
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Started | 133 | 133
Completed | 107 | 101
Not Completed | 26 | 32
Not completed — Death | 22 | 25
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery | Total
Number analyzed (Participants) | 133 | 133 | 266
Age, Continuous [Median (Full Range); unit: years] | 61 [26 to 81] | 61 [24 to 83] | 61 [24 to 83]
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 29 | 26 | 55
  51 - 65 years | 58 | 59 | 117
  > 65 years | 46 | 48 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 71 | 138
  Male | 66 | 62 | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
  United Kingdom | 16 | 10 | 26
  Spain | 1 | 1 | 2
  Canada | 13 | 15 | 28
  Netherlands | 10 | 11 | 21
  Sweden | 1 | 1 | 2
  Belgium | 1 | 5 | 6
  Norway | 6 | 7 | 13
  Denmark | 3 | 1 | 4
  Poland | 6 | 5 | 11
  Italy | 33 | 32 | 65
  France | 38 | 41 | 79
  Germany | 2 | 0 | 2
WHO performance status [Count of Participants; unit: Participants]
  PS 0: able to carry out all normal activity without restriction | 100 | 110 | 210
  PS 1: restricted in strenuous activity but ambulatory and able to carry out light work | 33 | 22 | 55
  PS 2: ambulatory and capable of all self-care but unable to carry out any work activities | 0 | 1 | 1
Concomitant non-malignant disease [Count of Participants; unit: Participants]
  No | 70 | 58 | 128
  Yes | 63 | 74 | 137
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Abdominal Recurrence or Death
Description: Abdominal recurrence was defined by one of the following events: local/abdominal or distant progressive disease during preoperative radiotherapy (as per RECIST 1.1), tumor or patient becoming inoperable (ASA score of 3 or involvement of superior mesenteric artery, aorta, or bone), peritoneal metastasis found at surgery, macroscopic residual disease left in at surgery (R2 resection), or local relapse (after macroscopically complete resection). Liver metastases were regarded as distant metastatic events. Patients with distant metastases were followed until local failure was detected. Patients without one of these events were censored at the date of last follow-up.
Time Frame: ARFS was measured from date of randomization to date of abdominal relapse or death, whichever occurred first, up to a maximum of 7 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 133 | 133
Participants
  No event | 72 | 73
  Event | 61 | 60
Statistical Analysis 1: Comparison: Surgery Alone vs Preoperative Radiotherapy Followed by En-bloc Surgery; Sample size was determined to provide 90% power for detecting a Hazard Ratio (HR)=0.52 (which corresponds to a 20% difference in ARFS rate at 5 years, from 50% in the surgery arm to 70% in the experimental arm) at a global 2-sided 5% significance level assuming ARFS followed an exponential distribution in both arms. This test required 102 events at the time of the statistical analysis; Test type: Superiority — Time assessment biases were taken into account for the primary endpoint: * Surgery alone arm: abdominal recurrence occurring prior to week 14 assessment was counted as occurring at week 14; progression occurring after the week 14 was counted as occurring at week 24. * Preoperative RT arm: abdominal recurrence occurring was counted as occurring at week 14; and any abdominal recurrence occurring after and prior to or during the week 24 will be counted as occurring at week 24; p = 0.955, Regression, Cox — A 5% significance level was considered as a threshold for statistical significance; The time assessment biases correction described before was not applied to patients for whom death was the first event; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.71 to 1.44] — The arm having surgery alone was the reference arm

2. Secondary Outcome: Acute Toxicity Profile of Preoperative Radiotherapy.
Description: The acute toxicity was assessed in randomized patients who received at least one dose of preoperative radiotherapy (RT). It follows Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 in the RT safety population, assuming the following classification:
  * Grade 0 No event reported
  * Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  * Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  * Grade 4 Life-threatening consequences; urgent intervention indicated.
  * Grade 5 Death related to AE. For each item of the CTCAE, the worst grade of acute toxicity from the data of randomization prior to surgery was taken
Time Frame: From date of randomization to the date of surgical procedure, prior to surgery
Population: Only patients in the "Preoperative radiotherapy followed by en-bloc surgery" that received at least one dose of radiotherapy were considered for this secondary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 0 | 127
Participants
  CTCAE Grade 0 |  | 4
  CTCAE Grade 1-2 |  | 106
  CTCAE Grade 3 |  | 15
  CTCAE Grade 4 |  | 1
  CTCAE Grade 5 |  | 1

3. Secondary Outcome: Perioperative Complications
Description: Adverse events and side effects possibly related to surgery were assessed according to the Dindo's classification. This scales the observed side effects as Grade 0 No event Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III Requiring surgical, endoscopic or radiological intervention Grade IV Life-threatening complication (including CNS complications) requiring IC/ICU-management Grade V Death of a patient For each item, the frequency of the worst grade of the observed toxicity was tabulated by treatment group.
  The perioperative period commence at the time of surgery (at the time of the induction anaesthesia) to the complete closure of the wound.
Time Frame: From the date of surgery, up to 60 days following surgery
Population: all randomized patients who are eligible and have started their allocated treatment (at least have been operated or received one fraction of irradiation followed by surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 128 | 119
Participants
  Dindo scale Grade 0 | 57 | 34
  Dindo scale Grade 1-2 | 57 | 58
  Dindo scale Grade 3 | 13 | 24
  Dindo scale Grade 4 | 1 | 2
  Dindo scale Grade 5 | 0 | 1

4. Secondary Outcome: Late Complications
Description: The late toxicities occurring more than 60 days after surgery. These were reported using Common Terminology Criteria for Adverse Events (CTCAE) v4.0. This scales the observed toxicity from Grade 1 to 5, assuming the following classification:
  * Grade 0 no event
  * Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  * Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  * Grade 4 Life-threatening consequences; urgent intervention indicated.
  * Grade 5 Death related to AE. Full AE reporting can be found in the Adverse Event Section.
Time Frame: From day 60 after surgery till end of follow-up, up to 7 years
Population: all randomized patients who are eligible and have started their allocated treatment (at least have been operated or received one fraction of irradiation)
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 128 | 127
Participants
  CTCAE Grade 0 | 58 | 53
  CTCAE Grade 1-2 | 51 | 50
  CTCAE Grade 3 | 17 | 20
  CTCAE Grade 4 | 2 | 4
  CTCAE Grade 5 | 0 | 0

5. Secondary Outcome: Tumor Response to Preoperative Radiotherapy
Description: For patients that received preoperative radiotherapy, the tumor response was assessed using RECIST 1.1. Response criteria were essentially based on a set of measurable lesions identified at baseline as target lesions, and followed at the end of the radiotherapy. Response was not the primary endpoint, so a confirmatory CT-scan was not mandatory.
Time Frame: Two weeks after completion of Pre-operative Radiotherapy, before Surgery
Population: Tumor response using RECIST 1.1 was only assessed for patients receiving preoperative radiotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 0 | 133
Participants
  Partial response |  | 4
  Stable disease |  | 99
  Progressive disease |  | 18
  Early death |  | 1
  Not evaluable |  | 11

6. Secondary Outcome: Number of Patients With an Abdominal Recurrence
Description: Abdominal recurrence was defined in the ARFS section. The following are considered competing events:
  * death in the absence of abdominal failure
  * distant metastases diagnosed before abdominal failure Patients without one of these events were censored at the date of last follow-up.
Time Frame: ARFI was measured from the date of randomization to the date of abdominal relapse, up to a maximum of 7 years
Population: Note that distant metastasis before or in the absence of abdominal recurrence was counted as a competing risk for this endpoint - whereas distant metastasis in the absence of abdominal recurrence was considered a non-event for the primary endpoint (ARFS). This explains the difference in non-events between the survival and interval endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 133 | 133
Participants
  No event (censored) | 61 | 65
  Abdominal recurrence | 46 | 48
  Competing event (see outcome measure description) | 26 | 20
Statistical Analysis 1: Comparison: Surgery Alone vs Preoperative Radiotherapy Followed by En-bloc Surgery; Test type: Superiority — ARFI was described using cumulative incidence curves. ARFI was compared between the two treatment arms using a Fine and Gray model; p = 0.658, Fine and Gray model — A 5% significance level was considered as a threshold for statistical significance; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.74 to 1.60]

7. Secondary Outcome: Number of Patients With Metastases or Death
Description: Alive and metastases free patients will be censored at the date of last follow-up.
Time Frame: Metastases free survival was measured from the date of randomization to the date of occurrence of distant metastases or death, whichever occurred first, up to a maximum of 7 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 133 | 133
Participants
  Alive and metastases free (censored) | 88 | 92
  metastasis and/or death (event) | 45 | 41
Statistical Analysis 1: Comparison: Surgery Alone vs Preoperative Radiotherapy Followed by En-bloc Surgery; Test type: Superiority; p = 0.595, Regression, Cox — A 5% significance level was considered as a threshold for statistical significance; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.58 to 1.36]

8. Secondary Outcome: Number of Patients Alive
Description: Alive patients were censored at the date of last follow-up. Causes of death were recorded and reported as a table.
Time Frame: Overall survival was measured from the date of randomization to the date of death, whatever the cause, up to a maximum of 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
Number analyzed (Participants) | 133 | 133
Participants
  Alive (censored) | 111 | 108
  Death (event) | 22 | 25
Statistical Analysis 1: Comparison: Surgery Alone vs Preoperative Radiotherapy Followed by En-bloc Surgery; Test type: Superiority; p = 0.615, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.65 to 2.05]

ADVERSE EVENTS:
Time Frame: Arm 1: within 21 days before randomization, 15 and 60 days after surgery, 14, 24, 36 and 48 weeks after randomization and (after week 48 after randomization) every 6 months until recurrence/death. Arm 2: within 21 days before randomization, weekly during the preoperative period, 2 weeks after end of RT, 15 days after surgery, 24 weeks after randomization, 60 days after surgery, 36 and 48 weeks after randomization and (after week 48 after randomization) every 6 months until recurrence/death.
Description: Patient population:
  * all cause mortality: all patients
  * serious and non-serious adverse events: safety population consisting of all randomized patients who are eligible and have started their allocated treatment (at least have been operated or received one fraction of irradiation)
Arm/Group | Surgery Alone | Preoperative Radiotherapy Followed by En-bloc Surgery
All-Cause Mortality (participants affected / at risk) | 22/133 | 25/133
Serious Adverse Events (participants affected / at risk) | 37/128 | 48/127
Other Adverse Events (participants affected / at risk) | 124/128 | 127/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Alone (N=128) | Preoperative Radiotherapy Followed by En-bloc Surgery (N=127)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (2)
ASCITES (Gastrointestinal disorders) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (2)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIAPHRAGMATIC HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (3)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTRIC FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROPLEURAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 3 (3)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 2 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 2 (2)
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 5 (6) | 5 (6)
JEJUNAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (3)
PANCREATIC FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 3 (5)
SUBILEUS (Gastrointestinal disorders) | 5 (5) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (3)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
ULCER (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEVICE OCCLUSION (Infections and infestations) | 0 (0) | 1 (1)
EMPYEMA (Infections and infestations) | 1 (1) | 0 (0)
GENITAL HERPES (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 1 (1)
PANCREATIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 2 (2) | 2 (2)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RETROPERITONEAL ABSCESS (Infections and infestations) | 3 (3) | 1 (1)
RETROPERITONEAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)
WOUND INFECTION (Infections and infestations) | 0 (0) | 2 (2)
ANASTOMOTIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA, OBSTRUCTIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PANCREATIC LEAK (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
PERIPANCREATIC FLUID COLLECTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 3 (3)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LARGE INTESTINE ANASTOMOSIS (Surgical and medical procedures) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 2 (3)
HAEMATOMA (Vascular disorders) | 2 (2) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 2 (2) | 1 (1)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1)
ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1)
LYMPHOCELE (Vascular disorders) | 0 (0) | 1 (1)
LYMPHORRHOEA (Vascular disorders) | 0 (0) | 1 (1)
NECROSIS ISCHAEMIC (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Alone (N=128) | Preoperative Radiotherapy Followed by En-bloc Surgery (N=127)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CAR OTH ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
CAR OTH TACHYCARDIA, PT ON CHEMOTHERAPY, NOT RELATED TO PRIMARY DISEASE TX (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 2 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 1 (3)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
END OTH PRECOCIOUS POSTMENOPAUSALITY (Endocrine disorders) | 0 (0) | 1 (1)
END OTH THYMIC HYPERPLASIA (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
EYE OTH AMAUROSIS FUGAX (Eye disorders) | 1 (1) | 0 (0)
EYE OTH CONJUNCTIVAL PALLOR (Eye disorders) | 0 (0) | 1 (1)
EYE OTH DIFFICULTY TO OPEN THE LEFT EYELID (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 (36) | 36 (74)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOATING (Gastrointestinal disorders) | 0 (0) | 3 (5)
BURN (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLONIC FISTULA (Gastrointestinal disorders) | 2 (2) | 1 (1)
COLONIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 11 (19) | 40 (83)
DIARRHEA (Gastrointestinal disorders) | 17 (29) | 59 (143)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 8 (10)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 4 (4)
GAS OTH ABDOMINAL CRAMPS (Gastrointestinal disorders) | 0 (0) | 2 (3)
GAS OTH ABDOMINAL METEORISM (Gastrointestinal disorders) | 0 (0) | 1 (2)
GAS OTH ABSCESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH ACCELERATION OF TRANSIT (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH BELCHING (Gastrointestinal disorders) | 1 (2) | 0 (0)
GAS OTH BOWEL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH COLON HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH DENTAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH DIGESIVE TROUBLE (IMPERIOSITY) (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH DIGESTIVE INTOLERANCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH DIGESTIVE TRANSIT (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH DIGESTIVE TROUBLE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH DIVERTICULITIS (MILD SYMPTOMS BUT NOT VISIBLE ON SCAN) (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH ENTERO-CUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (2)
GAS OTH ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH EPIGASTRIC PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2)
GAS OTH EXCACERBATION CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH FISTULOUS ORIFICE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH GASTRIC DISORDERS (Gastrointestinal disorders) | 0 (0) | 3 (3)
GAS OTH GASTRIC PAIN (Gastrointestinal disorders) | 0 (0) | 1 (3)
GAS OTH GASTROINTESTINAL DISORDERS (INTOLERANACE) (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH HEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH ILEAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH INCREASED URGENCY OF DEFECATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH INFECTED RETROPERITONEAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (2) | 0 (0)
GAS OTH INTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 0 (0) | 1 (2)
GAS OTH IVER COLIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH LEFT RETROPERITONEAL COLLECTION, POSSIBLE PANCREATIC LEAK (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH LOWER ABDOMINAL HEAVINESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH MALNUTRIRION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH OBSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH PAIN AT RIGHT HYPOCHONDRE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH PAIN AT RIGHT HYPOCONDRE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH POSTPRANDIAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH RETROPERITONEAL ABSCESS (Gastrointestinal disorders) | 1 (2) | 1 (1)
GAS OTH SENSITIVE ABDOMEN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH SUB-OCCLUSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH SUB-OCCLUSIVE SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH SUBOCLUSIVE SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS OTH SWELLING LEFT LOWER ABDOMEN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH TRANSIT DISORDERS (Gastrointestinal disorders) | 0 (0) | 2 (3)
GAS OTH TRANSIT TROUBLES (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAS OTH VAGUE ABDOMINAL COMPLAINTS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 2 (4) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 7 (15)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (4)
GASTROPARESIS (Gastrointestinal disorders) | 0 (0) | 2 (3)
ILEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 3 (4)
JEJUNAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 2 (5)
NAUSEA (Gastrointestinal disorders) | 10 (15) | 92 (333)
PANCREATIC FISTULA (Gastrointestinal disorders) | 1 (2) | 0 (0)
RECTAL FISTULA (Gastrointestinal disorders) | 0 (0) | 3 (3)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2)
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (3) | 2 (2)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2) | 29 (64)
CHILLS (General disorders) | 0 (0) | 1 (2)
EDEMA FACE (General disorders) | 0 (0) | 1 (1)
EDEMA LIMBS (General disorders) | 5 (9) | 12 (50)
EDEMA TRUNK (General disorders) | 0 (0) | 2 (6)
FATIGUE (General disorders) | 25 (41) | 91 (394)
FEVER (General disorders) | 2 (2) | 6 (7)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 1 (1)
GEN OTH ALTERATION OF THE GENERAL STATE (General disorders) | 0 (0) | 1 (2)
GEN OTH DISCRETE ACCELERATION OF TRANSIT (General disorders) | 0 (0) | 1 (1)
GEN OTH GENERAL STATUS IMPAIRMENT (General disorders) | 0 (0) | 1 (1)
GEN OTH NIGHT SWEATS (General disorders) | 0 (0) | 1 (1)
GEN OTH RADIATION PAIN (General disorders) | 0 (0) | 1 (3)
GEN OTH RIGHT SUB PUBIC PAIN (General disorders) | 0 (0) | 1 (1)
GEN OTH RIGHT SUS PUBIC PAIN (General disorders) | 0 (0) | 1 (1)
GEN OTH TRANSIT DISORDERS (General disorders) | 0 (0) | 1 (1)
GEN OTH WORSENING IN GENERAL CONDITION (General disorders) | 0 (0) | 1 (1)
LOCALIZED EDEMA (General disorders) | 1 (1) | 1 (1)
NECK PAIN (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (5)
PAIN (General disorders) | 12 (15) | 16 (50)
ALLERGIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BONE INFECTION (Infections and infestations) | 0 (0) | 1 (3)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 2 (2) | 2 (2)
INF OTH BLOOD INFECTION WITH STAPHYLOCOCCUS EPIDERMIS (Infections and infestations) | 1 (1) | 0 (0)
INF OTH CHEST INFECTION (Infections and infestations) | 0 (0) | 1 (4)
INF OTH CLOSTRIDIUM DIFFICILE (Infections and infestations) | 0 (0) | 1 (1)
INF OTH FUNGEMIA (Infections and infestations) | 0 (0) | 1 (1)
INF OTH HELICOBACTER PYLORI INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INF OTH HERPES GENITALIS (Infections and infestations) | 0 (0) | 1 (1)
INF OTH HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INF OTH HERPES ZOSTER IN RIGHT LUMBAR REGION ALMOST RESOLVED. (Infections and infestations) | 0 (0) | 1 (1)
INF OTH HERPES ZOSTER IN RIGHT LUMBAR REGION. (Infections and infestations) | 0 (0) | 1 (1)
INF OTH HSV-1 IN GENITAL AREA (Infections and infestations) | 0 (0) | 1 (1)
INF OTH INFECTED ABDOMINAL COLLECTION (Infections and infestations) | 0 (0) | 1 (1)
INF OTH INFECTED POST-OPERATIVE COLLECTION (Infections and infestations) | 0 (0) | 1 (1)
INF OTH SURGICAL BED INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1)
INF OTH UNSPECIFIC INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INF OTH ZONA (Infections and infestations) | 0 (0) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 1 (2)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 2 (4)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 6 (7)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (1) | 30 (63)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH DIAFRAGMATIC HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH EVENTRATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
INJ OTH EVENTRATION SURGERY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 4 (11) | 1 (1)
INJ OTH INTESTINAL ADHESIONS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH LEFT INGUINAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH RETROPERITONEAL FLUID COLLECTION (NEGATIVE FOR INFECTION) (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
INJ OTH RIGHT INGUINAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH SMALL RETROPERITONEAL COLLECTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH SURGERY WOUND SENSITIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJ OTH WOUND PAIN (INTERMITTENT) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INJ OTH WOUND SURGERY PAINFUL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (5)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 3 (5) | 2 (4)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 5 (10) | 5 (10)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0)
CPK INCREASED (Investigations) | 1 (1) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (2) | 0 (0)
INR INCREASED (Investigations) | 1 (1) | 0 (0)
INV OTH DECREASED IRON (Investigations) | 0 (0) | 1 (1)
INV OTH INFLAMMATORY SYNDROME (Investigations) | 0 (0) | 1 (1)
INV OTH LDH INCREASED (Investigations) | 1 (1) | 0 (0)
INV OTH URINE OUTPUT INCREASED (Investigations) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 5 (20) | 4 (7)
WEIGHT LOSS (Investigations) | 23 (41) | 63 (160)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 11 (14) | 61 (160)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (5) | 5 (6)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (7) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
MET OTH MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 18 (30)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 12 (25)
MUS OTH ARTICULAR PAIN AT LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH DORSAL ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH INGUINAL HERNIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH INGUINLA HERNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH LEFT ILIAC FOSSA ABSCESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH LEFT LIMB MUSUCLAR DEFICIT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MUS OTH LUMBAR FOSSA MUSCULAR CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH MASTICATION PROBLEM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH MUSCLE CRAMPS LEGS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH MUSCULAR CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PAIN (LUMBAR REGION) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PAIN AND MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PAIN AND MUSCLES CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PAIN AT THE LEFT LEG (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
MUS OTH PAIN AT THE LEFT LUMBAR FOSSA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PAIN AT THIGH (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH PARAVERTEBRAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH RIGHT INGUINAL HERNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
MUS OTH RIGHT LUMBAR FOSSA PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH RIGHT PARAVERTEBRAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH RIGHT SHOULDER AND RIGHT SIRLOIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH SHOULDER PAIN (LEFT) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUS OTH SURGERY WOUND SENSATIVE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
MUS OTH TENDON RUPTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUS OTH TRUNK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS TRUNK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (7)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEO OTH GASTRIC POLYP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (9)
DIZZINESS (Nervous system disorders) | 1 (1) | 3 (3)
DYSESTHESIA (Nervous system disorders) | 3 (4) | 4 (7)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 6 (8)
HEADACHE (Nervous system disorders) | 5 (7) | 14 (26)
ISCHEMIA CEREBROVASCULAR (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH CRURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH DEAFFERENTATION PAIN (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH HYPERSENSITIVITY OF THE EXTERNAL FACE OF THE RIGHT THIGH (Nervous system disorders) | 0 (0) | 1 (2)
NER OTH INSENSIBILITY PART RIGHT HIP (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH ISCHEMIC INFARCTION BRAIN (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH L5 DISTAL DEFICIT (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH LEFT GROIN/THIGH NUMBNESS (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH LEG NUMBNESS (LEFT) (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH LEG NUMBNESS (LEG) (Nervous system disorders) | 1 (1) | 0 (0)
NER OTH NEUROGENIC PAIN (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH NEUROPATHIC PAIN (Nervous system disorders) | 1 (6) | 0 (0)
NER OTH NUMBNESS (LEFT THIGH) (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH NUMBNESS LEFT LEG (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH NUMBNESS LEFT THIGH (Nervous system disorders) | 1 (3) | 0 (0)
NER OTH NUMBNESS RIGHT LEG (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH PARAPLEGIA (Nervous system disorders) | 1 (7) | 0 (0)
NER OTH RIGHT BIG TOE HYPOESTHESIA (Nervous system disorders) | 1 (2) | 0 (0)
NER OTH RIGHT SCIATICA (Nervous system disorders) | 0 (0) | 1 (2)
NER OTH SENSITIVITY TO THE LOWER PART OF THE STERNUM (Nervous system disorders) | 1 (1) | 0 (0)
NER OTH SENSORY DEFICIT AT THE ANTERIOR FACE OF THE LEFT THIGH (Nervous system disorders) | 0 (0) | 1 (1)
NER OTH SEQUELAE AFTER ISCHEMIC INFARCTION BRAIN (Nervous system disorders) | 0 (0) | 1 (2)
NER OTH SPONGY FEELING LEFT FOSSA ILIACA (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 3 (3)
PARESTHESIA (Nervous system disorders) | 6 (16) | 5 (5)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 6 (13) | 3 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 14 (30) | 15 (24)
STROKE (Nervous system disorders) | 2 (2) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
VASOVAGAL REACTION (Nervous system disorders) | 1 (1) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 4 (7)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 3 (4)
DEPRESSION (Psychiatric disorders) | 1 (1) | 4 (6)
INSOMNIA (Psychiatric disorders) | 0 (0) | 3 (6)
PSY OTH SLEEP DISORDERS (Psychiatric disorders) | 1 (1) | 1 (2)
PSY OTH SOCIAL PHOBIA (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (2)
ADRENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 3 (4) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 2 (2)
REN OTH ACUTE RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH BASELINE URINARY SYMPTOMS, OTHER. (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH BLADDER LITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH BLOCKED URINARY CATHETER (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH INGUINAL HERNIA (Renal and urinary disorders) | 0 (0) | 1 (1)
REN OTH POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
REN OTH RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0)
REN OTH RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (2) | 2 (2)
REN OTH SYNDROME OF JUNCTION OF THE LEFT KIDNEY (Renal and urinary disorders) | 1 (2) | 0 (0)
REN OTH URINARY DISORDERS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1) | 5 (9)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 3 (3) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 1 (2)
EJACULATION DISORDER (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (8) | 0 (0)
GENITAL EDEMA (Reproductive system and breast disorders) | 3 (7) | 1 (1)
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PREMATURE MENOPAUSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
REP OTH HYDROCELE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
REP OTH RIGHT SIDE VARICOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
REP OTH TESTICULAR OEDEMA (LEFT) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
SCROTAL PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 2 (3) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (13)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH BIBASAL INSPIRATORY CRACKLES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH BREATHLESSNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
RES OTH COPD (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
RES OTH EMPYEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RES OTH PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH PULMONARY EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RES OTH RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH RIGNT POSTERIOR PARIETAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RES OTH SHORTNESS OF BREATH, PT ON CHEMO, NOT RELATED TO PRIMARY DISEASE TX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RES OTH THORACIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH EPITHELITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH CUTANEOUS ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH EPITHELITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
SKI OTH HYPERSENSITIVITY SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH ITCHING AREA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH KELOID SCAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKI OTH PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKI OTH RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH SCAR HYPERTROPHIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKI OTH SKIN AND SUBCUTANEOUS TISSUE (FOLLICULITIS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKI OTH SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKI OTH TOXICODERMIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN INFECTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 2 (2) | 0 (0)
HOT FLASHES (Vascular disorders) | 0 (0) | 1 (2)
HYPERTENSION (Vascular disorders) | 10 (24) | 10 (30)
HYPOTENSION (Vascular disorders) | 4 (4) | 5 (9)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2) | 7 (24)
VAS OTH AORTIC ECTASIA (Vascular disorders) | 1 (1) | 0 (0)
VAS OTH INFERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 1 (9)
VAS OTH PULMONARY EMBOLISM (Vascular disorders) | 1 (5) | 0 (0)
VASCULITIS (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial is limited by the short follow-up. An update will be done in 5 years. The trial is not powered for a difference in survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT01344018/Prot_SAP_000.pdf